CLINICAL TRIAL: NCT05538585
Title: A Food-Effect Study for the Safety and Assessment of Pharmacokinetics of Navocaftor and Galicaftor.
Brief Title: A Study to Assess How Food Affects the Safety and Pharmacokinetics of Galicaftor and Navocaftor
Acronym: M23-492 FE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M23-492
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: Galicaftor; Navicaftor; ABBV-3067; ABBV-2222
MeSH Terms: interventions — GLPG2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: Navocaftor with food (Experimental): Participants will receive navocaftor administered with food
  Interventions: Drug: Navocaftor
- Part 1: Navocaftor without food (Experimental): Participants will receive navocaftor administered without food
  Interventions: Drug: Navocaftor
- Part 2: Galicaftor with food (Experimental): Participants will receive galicaftor administered with food
  Interventions: Drug: Galicaftor
- Part 2: Galicaftor without food (Experimental): Participants will receive galicaftor administered without food
  Interventions: Drug: Galicaftor

INTERVENTIONS:
Drug: Galicaftor — Oral
  Other Names: ABBV-2222
  Arms: Part 2: Galicaftor with food; Part 2: Galicaftor without food
Drug: Navocaftor — Oral
  Other Names: ABBV-3067
  Arms: Part 1: Navocaftor with food; Part 1: Navocaftor without food

SUMMARY:
Cystic Fibrosis (CF) is a rare, life-threatening, genetic disease that affects the lungs and digestive system, significantly impairing the quality of life, with those affected having a median age of death at 40. The objectives of this study are to assess the effect of food on the safety and pharmacokinetics of navocaftor and galicaftor.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is => 18.0 to <= 32.0 kg/ m2 after rounding to the tenth's decimal.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic, or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection, etc.].
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 4
  Cmax will be assessed.
Time to Cmax (peak time, Tmax) | Up to Day 4
  Tmax will be assessed.
Terminal Elimination Half-life (t1/2) | Up to Day 4
  Terminal elimination half-life (t1/2) will be assessed.
Area under the plasma curve (AUC) | Up to Day 4
  AUC will be assessed.
Number of Participants with Adverse Events (AEs) | Up to Day 38
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami /ID# 249531, Miami, Florida
  - Acpru /Id# 249532, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.abbvieclinicaltrials.com/study/?id=M23-492